CLINICAL TRIAL: NCT01092884
Title: Polypodium Leucotomos Extract as an Adjunct to Sunscreen for the Treatment of Melasma
Brief Title: Polypodium Leucotomos Extract for the Treatment of Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Industrial Farmacéutica Cantabria, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 092009-036
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2010-03

CONDITIONS: Melasma
Keywords: melasma; sunscreen; polypodium leucotomos
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Polypodium leucotomos (Active Comparator): Subjects randomized to this arm will receive oral supplementation with Polypodium leucotomos extract
  Interventions: Dietary Supplement: Polypodium leucotomos extract
- Sugar pill (Placebo Comparator): Subjects randomized to this arm will receive oral supplementation with placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Polypodium leucotomos extract — 240 mg capsule of Polypodium leucotomos extract will be taken orally three times daily
  Other Names: Heliocare
  Arms: Polypodium leucotomos
Other: Placebo — This placebo capsule will be taken orally three times daily
  Arms: Sugar pill

SUMMARY:
We will assess whether oral supplementation with Polypodium leucotomos, a commercially marketed fern extract, improves facial melasma in Hispanic women with moderate to severe melasma. Subjects will be randomized to either Group 1, which will receive oral Polypodium leucotomos extract plus topical sunscreen, or Group 2, which will receive oral placebo plus topical sunscreen. The study will last 12 weeks, and we hypothesize that the Polypodium leucotomos group will have more improvement in their melasma compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic female with moderate to severe facial melasma

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Recent use of hydroquinone, topical retinoids, topical steroids, or mechanically abrading procedures (such as laser therapy or dermabrasion) to the face
* Frequent use of tanning parlors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Mexameter score | 12 weeks
  Using rapid, non-invasive, narrow-band reflectance spectrophotometry (Mexameter), we will assess change in intensity of pigment in affected skin versus unaffected skin at 12 weeks

SECONDARY OUTCOMES:
MASI Score | 12 weeks
  We will use the standardized Melasma Area and Severity Index (MASI) score, assessed by blinded physician investigator, to assess change in severity of melasma at 12 weeks compared to baseline
Melasma-Related Quality of Life | 12 weeks
  We will use a validated questionnaire tool to assess change in melasma-related quality of life at 12 weeks compared to baseline